CLINICAL TRIAL: NCT03241511
Title: Pilot and Feasibility Clinical Research Grants in Kidney or Urologic Diseases (R21)
Brief Title: Novel PAradigm to Improve Inflammatory Burden in ESRD (rePAIR): A Pilot and Feasibility Randomized Controlled Trial
Acronym: rePAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-111-1; R21DK108076 (NIH)
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Chronic Periodontitis; End Stage Renal Disease
Keywords: Periodontitis, End Stage Renal Disease, Periodontal treatment
MeSH Terms: conditions — Chronic Periodontitis; Kidney Failure, Chronic; Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Briefly, treatment sessions will include oral hygiene behavioral modification and scaling and root planning (removing the bacterial biofilm and calculus below the gum line) in order to eliminate etiologic factors and control periodontal inflammation. Once the treatment sessions are completed, the patients will enter the maintenance phase and will be followed for 6 months. In this phase, the patients will receive systematic and repeated supportive periodontal treatment (tooth cleanings above the gum line with re-enforcement of oral hygiene). Outcomes will be assessed at 2-, 4-, and 6-months. Throughout the course of the study, additional dental needs will be addressed with immediate referral to the subject's general dentist or clinics at the University of Connecticut.
  Interventions: Other: Test
- Control (No Intervention): The Control arm will receive only a single treatment session without maintenance sessions (see visit Table in Human Subject Protection section). Outcomes will be assessed at 2-, 4-, and 6-months.

INTERVENTIONS:
Other: Test — Briefly, treatment sessions will include oral hygiene behavioral modification and scaling and root planning (removing the bacterial biofilm and calculus below the gum line) in order to eliminate etiologic factors and control periodontal inflammation. Once the treatment sessions are completed, the patients will enter the maintenance phase and will be followed for 6 months. In this phase, the patients will receive systematic supportive periodontal treatment (tooth cleanings above the gum line with re-enforcement of oral hygiene).
  Arms: Test

SUMMARY:
The goal of this project is to assess repeated and ongoing oral care and the way it may affect inflammation and quality of life in hemodialysis patients. Two treatment groups will be compared:

* 1) ongoing and repeated gum disease therapy including deep tooth cleaning followed by multiple appointments of maintenance
* 2) single session of gum disease therapy with only one session of deep tooth cleaning Samples of blood will be obtained for study to examine the changes of inflammatory substances in the blood as a result of the two different gum disease treatments. Also, a 14-question survey will be discussed with you to assess oral health related quality of life (OHIP-14) and the way it is affected by oral care.

For this project, four dialysis centers will be randomly assigned to either of the treatment groups #1 or #2 prior to your enrollment. For this purpose, there are two distinct consent forms explaining the visits, procedures and risks of the two treatment groups #1 or #2. As a result, all participants in the same dialysis center will belong to the same treatment group (either #1 or #2) and presented with the corresponding consent form.

This dialysis center has been randomized to treatment group # 1; therefore you will receive ongoing and repeated gum disease therapy including deep tooth cleaning followed by multiple appointments of maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be referred by nephrologist
* Patient must be diagnosed with ESRD and on Hemodialysis
* life expectancy more than one year
* at least 21 years of age
* 12 or more teeth
* must meet the Periodontal diagnosis criteria (The diagnosis of periodontitis is based on the definition of moderate periodontitis with at least 2 sites with CAL≥4mm or at least 2 sites with PD≥5mm not on the same tooth (Page and Eke 2007).)

Exclusion Criteria:

* Anticipating a kidney transplant
* AIDS
* Active malignancy
* Poor adherence to hemodialysis
* Dementia
* Currently prescribed anti-inflammatory medication
* Temporary catheter for dialysis access
* Gum disease treatment within the last year

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Serum CRP | 6 months
  Inflammatory markers

SECONDARY OUTCOMES:
Probing depth PD | 6 months
  Clinical periodontal outcome
Clinical attachment levels CAL | 6 months
  Clinical periodontal outcome
OHIP-14 | 6 months
  Patient Centered Outcome
Serum IL-6 | 6 months
  Inflammatory Marker
F2 isoprostanes | 6 months
  Oxidative Stress Marker
isofurans | 6 months
  Oxidative Stress Marker

CONTACTS AND LOCATIONS:
Overall Officials: Effie Ioannidou, DDS, MS, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the study is completed, the data will be available without cost to researchers. As part of the registration process, users must agree to the conditions of use governing access to the public release data (e.g., data destruction after analyses are complete, proper acknowledgement of data resources). Data will be provided at no cost and all data will be de-identified prior to sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will available after the completion of the study
Access Criteria: As part of the registration process, users must agree to the conditions of use governing access to the public release data (e.g., data destruction after analyses are complete, proper acknowledgement of data resources). Data will be provided at no cost and all data will be de-identified prior to sharing.

REFERENCES:
- [Background] Trivedi R, Fares G, Nunez VB, Campbell R, Clement M, Burleson J, Himmelfarb J, Ioannidou E. Novel PAradigm to improve Inflammatory burden in end stage Renal disease (rePAIR): study protocol for a randomized controlled trial. Trials. 2018 Jul 11;19(1):370. doi: 10.1186/s13063-018-2760-y. PMID 29996883

DOCUMENTS (1):
  • Study Protocol (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT03241511/Prot_000.pdf